CLINICAL TRIAL: NCT00166270
Title: Post Approval Study: MR Guided Focused Ultrasound Surgery in the Treatment of Uterine Fibroids
Brief Title: MR Guided Focused Ultrasound Surgery in the Treatment of Uterine Fibroids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UF014
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2018-07-09 (Actual); Status verified 2018-07

CONDITIONS: Uterine Fibroids
Keywords: Fibroids; ExAblate; MrgFus; Uterine Fibroids
MeSH Terms: conditions — Leiomyoma

ARMS (1):
- 1 (Experimental)
  Interventions: Device: ExAblate 2000

INTERVENTIONS:
Device: ExAblate 2000

SUMMARY:
This is a prospective, nonrandomized, multi-center study to evaluate the safety and effectiveness of ExAblate in the treatment of uterine fibroids. All patients will be treated and then followed for 36 months to evaluate the change in their fibroid symptoms.

DETAILED DESCRIPTION:
After the PMA Panel, the sponsor was requested to conduct a post-approval study. The objective of this study is to gather additional data to evaluate the safety and long term effectiveness of focused ultrasound treatment, and to include a larger cohort of African-American patients. Patients will be treated following the approved commercial treatment guidelines.

Uterine leiomyoma (fibroids) are the most common neoplasms of the female pelvis. These benign tumors are generally oval in shape, and often highly vascular. On T2 weighted MR imaging exams, or T1 exams with contrast, uterine fibroids are easily identifiable. They occur in 20-25% of women of reproductive age and can cause a variety of problems generally described as either bleeding or mass effects from the fibroid. In general, these symptoms can be classified into two categories:

1. heavy menstrual bleeding, defined as bleeding on heavy days requiring a change of sanitary wear every 2 hours or less, significant clot passage, flooding, substantial prolongation of menstrual periods compared with the patient's prior experience, or anemia.
2. pelvic pain or pressure, heaviness or discomfort, or similar symptoms in the back, flank or leg attributable to the bulk of the fibroid, urinary frequency, increase in nocturia, difficulty voiding or compression of the ureters with hydronephrosis.

Measures of the clinical success of patients who elect treatment of fibroids are generally subjective, and evaluated by the patient in terms of improvement in the initial symptoms that caused her to seek treatment (decrease in pain, bladder or bowel symptoms, or reduction in vaginal bleeding), while experiencing a minimum of co-morbidities from the treatment itself.

ELIGIBILITY:
Inclusion Criteria:

* Women who present with symptomatic uterine fibroids and are not seeking treatment for the reason of improving fertility.
* Able and willing to give consent and able to attend all study visits.
* Patient is pre or peri-menopausal (within 12 months of last menstrual period).
* Able to communicate sensations during the ExAblate procedure.
* Uterine fibroids, which are device accessible (i.e., positioned in the uterus such that they can be accessed without being shielded by bowel or bone).
* Fibroids(s) clearly visible on non-contrast MRI.

Exclusion Criteria:

* Metallic implants that are incompatible with MRI
* Sensitive to MRI contrast agents
* Severe claustrophobia that would prevent completion of procedure in MR unit
* Who are pregnant or desire to become pregnant in the future. Pregnancies following ExAblate treatment could be dangerous for both mother and fetus.
* Pedunculated fibroids
* Active pelvic inflammatory disease (PID)
* Active local or systemic infection
* Known or suspected pelvic carcinoma or pre-malignant conditions, including sarcoma and adenomatous hyperplasia
* Intrauterine device (IUD) anywhere in the treatment path
* Dermoid cyst of the ovary anywhere in the treatment path
* Extensive abdominal scarring that cannot be avoided by redirection of the beam (e.g., due to Caesarean section or repeated abdominal surgeries)
* Undiagnosed vaginal bleeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2005-01; Primary Completion 2006-04 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Measures of the clinical success of patients who elect treatment of fibroids are generally subjective, and evaluated by the patient in terms of improvement. | Within 1 month of Treatment

CONTACTS AND LOCATIONS:
Overall Officials: Phyllis Gee, M.D., Principal Investigator — North Texas UFI; Paul Curtis, M.D., Principal Investigator — Virtua; George Holland, M.D., Principal Investigator — Lahey Clinic; Dennis Sarti, M.D., Principal Investigator — Radnet Management; Fred Steinberg, M.D., Principal Investigator — Univeristy MRI; Elizabeth Stewart, M.D., Principal Investigator — Brigham and Women's Hospital
Locations (6):
- United States (6):
  - Radnet Management, Los Angeles, California
  - University MRI, Boca Raton, Florida
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Lahey Clinic, Burlington, Massachusetts
  - Virtua, Voorhees Township, New Jersey
  - North Texas Uterine Fibroid Institute, Plano, Texas

REFERENCES:
- See also: Sponsor web page — http://www.insightec.com